CLINICAL TRIAL: NCT03883607
Title: An Open Label, Randomized, Multicenter Study to Assess the Pharmacokinetic and Pharmacodynamic Profile and the Safety and Tolerability of Two Dose Levels of Elafibranor (80 mg and 120 mg) in Children and Adolescents, 8 to 17 Years of Age, With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Elafibranor, PK and Safety in Children and Adolescents 8 to 17 Years of Age With Non Alcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of efficacy (but not due to safety) in a Phase 3 trial of elafibranor in adult participants with NASH and fibrosis, this study in pediatric NASH was prematurely terminated
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFT505E-218-1; 2019-003400-12 (EudraCT Number)
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: Pediatric; Pharmacokinetics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elafibranor 80 mg (Experimental): Participants received Elafibranor 80 mg tablet orally once daily for 12 weeks.
  Interventions: Drug: Elafibranor 80mg
- Elafibranor 120 mg (Experimental): Participants received Elafibranor 120 mg tablet orally once daily for 12 weeks.
  Interventions: Drug: Elafibranor 120mg

INTERVENTIONS:
Drug: Elafibranor 80mg — Once daily oral intake of elafibranor 80 mg during 3 months
  Other Names: GFT505
  Arms: Elafibranor 80 mg
Drug: Elafibranor 120mg — Once daily oral intake of elafibranor 120 mg during 3 months
  Other Names: GFT505
  Arms: Elafibranor 120 mg

SUMMARY:
The study was being conducted in order to assess the pharmacokinetics and the safety of elafibranor following once daily administration of two dose levels of elafibranor (80 milligrams [mg] and 120mg) during 3 months in children and adolescent population (8 to 17 years of age) with non alcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Was male or female between 8 and 17 years of age (inclusive) at the time of Screening Visit (when consent for study participation is given) and at the time of Randomization;
* Diagnosis of NASH confirmed by histological evaluation (with or without fibrosis) from a liver biopsy obtained within 24 months prior to Randomization;
* Had an alanine aminotransferase (ALT) level greater than (>) 50 international units per liter (IU/L), at Screening;
* Had a Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) greater than or equal to (>=) 5, at Screening;
* Had a Body Mass Index z-score (BMI z-score) (also referred to as BMI-for-age percentile) >=85th percentile for age and gender at Screening;
* Had a Hemoglobin A1C (HbA1c) less than or equal (<=) to 8.5%. If the participants had Type 2 diabetes and is taking anti-diabetic therapy (e.g., metformin or insulin), treatment must had been started at least 3 months prior to Screening and the dose must had been stable for at least 3 months prior to Screening and should remain stable through Randomization;
* Sexually active female participants of childbearing potential must had agree to utilize a highly effective method of contraception per the Clinical Trial Facilitation Group Guidelines from Screening through 30 days after the last dose of study drug (1 month after the end of treatment), and agree to monthly pregnancy testing during the study up to and including end of study.

Other inclusion criteria may apply

Exclusion Criteria:

* Had history of bariatric surgery or planned surgery during the study period;
* Had known history of heart disease;
* Had uncontrolled hypertension evidenced by sustained elevation in systolic blood pressure greater than140 mmHg or diastolic blood pressure greater than 90 mmHg despite treatment with antihypertensive therapy, prior to Randomization;
* Had a known history of Type 1 diabetes;
* Had a known history of acquired immunodeficiency syndrome or positive screening for human immunodeficiency virus antibodies at Screening Visit;
* Had a documented weight loss of more than 5% during the 6-month period prior to Randomization;
* Had a history of renal disease defined as an estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m^2 using the Schwartz Bedside GFR Calculator for Children or present at Screening Visit;
* History of, significant alcohol consumption or inability to reliably quantify alcohol intake, and/or use of illicit drugs.
* Had clinical and/or historical evidence of cirrhosis, included by not limited to:

  1. Abnormal hemoglobin (with the exception of females with a documented history of a low hemoglobin during menstruation);
  2. White blood cell count less than 3,500 cells/mm^3 of blood;
  3. Platelet count less than150,000 cells/mm^3 of blood;
  4. Direct bilirubin greater than 0.3 mg/dL;
  5. Total bilirubin greater than 1.3 mg/dL unless the patient has a diagnosis of Gilbert disease in which case direct bilirubin, reticulocyte count and haemoglobin must be normal;
  6. Serum albumin less than 3.5 g/dL;
  7. International normalized ratio (INR) greater than 1.4;
* Has evidence of chronic liver disease other than NASH, defined by any one of the following:

  1. Biopsy consistent with histological evidence of autoimmune hepatitis;
  2. Serum hepatitis A antibody positive;
  3. Serum hepatitis B surface antigen positive;
  4. Serum hepatitis C antibody positive;
  5. Serum hepatitis E antibody positive;
  6. History of or current positive Anti-Mitochondrial Antibody Test;
  7. Known or current Iron/total iron binding capacity ratio (transferrin saturation) greater than 45% with histological evidence of iron overload;
  8. Known or current Alpha-1-antitrypsin phenotype/genotype ZZ or SZ;
  9. Diagnosis of Wilson's disease;
* Had AST and/or ALT greater than 8 fold the upper limit of normal;
* Was pregnant, lactating or is planning to become pregnant during the study;

Other exclusion criteria may apply

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Addy, MD MMSc, Study Director — Genfit
Locations (2):
- United States (2):
  - University of California, San Diego, California
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goyal NP, Mencin A, Newton KP, Durelle J, Carrier C, Ugalde-Nicalo P, Noel B, Mouton J, Vargas D, Magrez D, Tadde B, Birman P, Best BM, Addy C, Schwimmer JB. An Open Label, Randomized, Multicenter Study of Elafibranor in Children With Nonalcoholic Steatohepatitis. J Pediatr Gastroenterol Nutr. 2023 Aug 1;77(2):160-165. doi: 10.1097/MPG.0000000000003796. Epub 2023 Apr 21. PMID 37084342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 centers in the United Sates from 25 June 2019 and 16 June 2020. A total of 27 participants were screened, of which 10 participants were enrolled and randomized (1:1 ratio) to receive elafibranor 80 milligrams (mg)/120 mg sequentially. A total of 17 participants failed screening mainly due to not meeting eligibility criteria.
Pre-assignment Details: Screening was performed up to 4 weeks before study drug administered. Randomization was stratified by age (Cohort 1: greater than or equal to [>=] 12 to less than or equal to [<=] 17 years of age and Cohort 2: >=8 to <=11 years of age) and participant's historical fibrosis severity stage (stratum 1: fibrosis stage 0 to 1 and stratum 2: fibrosis stage 2 to 3). Due to lack of efficacy study was prematurely terminated, only Cohort 1 participants were involved in this study.
Groups:
- Elafibranor 80 mg: Participants received Elafibranor 80 mg tablets orally once daily for 12 weeks.
- Elafibranor 120 mg: Participants received Elafibranor 120 mg tablets orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Started (Randomized and treated participants.) | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population that had included participants who were randomized and had received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.52 (2.23) | 15.70 (2.31) | 15.11 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Elafibranor and Its Active Metabolite (GFT1007)
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Day 1: at pre-dose; Day 29: at pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours post dose; Day 30 and 85: at 24 hours after previous day dose administration
Population: Analysis was performed on PK population that included all participants who had received at least 1 dose of the study drug, did not had protocol deviations or adverse events (AEs) that significantly affected the PK, and had at least 1 post-dose PK sample.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
nanograms per milliliter (ng/mL)
  Elafibranor | 385.216 (218.646) | 658.054 (403.201)
  GFT1007 | 2367.620 (1088.123) | 2875.280 (1443.324)

2. Primary Outcome: Pharmacokinetics: Time to Maximum Observed Plasma Concentration (Tmax) of Elafibranor and Active Metabolite (GFT1007)
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
hours
  Elafibranor | 1.50 [0.52 to 2.00] | 1.00 [0.98 to 1.50]
  GFT1007 | 2.00 [1.50 to 2.00] | 1.50 [1.00 to 1.50]

3. Primary Outcome: Pharmacokinetics: Area Under The Plasma Concentration-time Curve From 0 to 24 Hours (AUC0-24) of Elafibranor and Active Metabolite (GFT1007)
Description: AUC0-24 defined as the area under the plasma concentration versus time curve of the study drug from time 0 to 24 hours.
Time Frame: as for outcome 1
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
nanograms*hour per milliliter
  Elafibranor | 973.301 (311.803) | 1457.728 (724.018)
  GFT1007 | 10011.405 (3575.220) | 10532.930 (3257.220)

4. Primary Outcome: Pharmacokinetics: Terminal Elimination Half-life ( t½) of Elafibranor and Active Metabolite (GFT1007)
Description: Plasma t1/2 was defined as the time taken by drug to reduce to half of its initial plasma concentration.
Time Frame: as for outcome 1
Population: Analysis was performed on PK population. Here, 'number analyzed' signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
hours
  Elafibranor: number analyzed (Participants) | 1 | 3
  Elafibranor | 34.170 (NA) — Since one participant was evaluated, standard deviation (SD) was not calculable. | 37.620 (15.473)
  GFT1007: number analyzed (Participants) | 4 | 5
  GFT1007 | 9.572 (5.592) | 6.682 (1.120)

5. Primary Outcome: Pharmacokinetics: Plasma Trough Concentrations (Ctrough) of Elafibranor and Active Metabolite (GFT1007)
Description: Ctrough was defined as the plasma concentration of study drug observed just before treatment administration during repeated dosing.
Time Frame: Pre-dose on Day 1 and 29
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
ng/mL
  Elafibranor | 14.904 (3.516) | 29.035 (15.087)
  GFT1007 | 97.771 (49.636) | 55.243 (27.769)

6. Secondary Outcome: Pharmacodynamics (PD) - Liver Markers: Change From Baseline in Serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT), and Alkaline Phosphatase (ALP) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1. Missing data were not imputed for the analysis. Normal range at screening: AST: 0 - 39 international units per liter (IU/L), ALT: 5 - 30 IU/L, GGT: 2 - 24 IU/L, and ALP: 74 - 390 IU/L.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: Analysis was performed on ITT population. Here, 'number analyzed' signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
IU/L
  ALT: Day 15 | 4.2 (21.7) | -13.8 (25.0)
  ALT: Day 29 | -0.2 (35.9) | -27.6 (18.4)
  ALT: Day 57 | 0.2 (27.3) | -30.8 (16.5)
  ALT: Day 85 | 17.8 (56.6) | -34.6 (25.6)
  ALT: Day 113: number analyzed (Participants) | 4 | 4
  ALT: Day 113 | 37.3 (46.9) | -28.0 (22.2)
  AST: Day 15 | 4.0 (16.0) | 0.8 (9.5)
  AST: Day 29 | 4.0 (16.3) | -4.0 (9.5)
  AST: Day 57 | 1.0 (6.1) | -5.8 (4.1)
  AST: Day 85 | 7.4 (15.3) | -8.2 (8.3)
  AST: Day 113: number analyzed (Participants) | 4 | 4
  AST: Day 113 | 9.3 (8.4) | -7.8 (8.7)
  GGT: Day 15 | -9.2 (6.8) | -8.8 (4.4)
  GGT: Day 29 | -15.6 (9.9) | -16.0 (5.9)
  GGT: Day 57 | -1.0 (20.7) | -15.6 (9.1)
  GGT: Day 85 | 11.2 (39.1) | -16.2 (9.9)
  GGT: Day 113: number analyzed (Participants) | 4 | 4
  GGT: Day 113 | 45.3 (43.8) | -9.5 (6.6)
  ALP: Day 15 | -4.6 (23.1) | -18.0 (11.2)
  ALP: Day 29 | -24.8 (28.4) | -14.6 (8.1)
  ALP: Day 57 | -28.2 (36.5) | -18.4 (8.2)
  ALP: Day 85 | -32.6 (51.5) | -25.0 (12.4)
  ALP: Day 113: number analyzed (Participants) | 4 | 4
  ALP: Day 113 | -7.8 (45.4) | -16.8 (10.2)

7. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Adiponectin at Days 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1. Missing data were not imputed for the analysis.
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: Analysis was performed on ITT population. Here, 'number analyzed' signifies participants who were evaluable for this outcome measure at the specific timepoints.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
micrograms per milliliter (mcg/mL)
  Day 29 | 0.2410 (0.3729) | 0.2112 (1.0304)
  Day 57 | 0.5780 (1.0530) | -0.2752 (1.0022)
  Day 85 | 0.3372 (1.4844) | -0.0590 (1.0476)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | -0.4663 (0.8972) | 0.0322 (1.0588)

8. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Cytokeratin 18 (CK-18)/M65 and CK-18/M30 at Days 29, 57, 85, and 113
Description: as for outcome 7
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
IU/L
  CK-18/M65: Day 29 | 39.412 (346.370) | -70.902 (121.905)
  CK-18/M65: Day 57 | -30.302 (326.632) | -60.578 (186.165)
  CK-18/M65: Day 85 | -2.320 (231.775) | -122.070 (265.059)
  CK-18/M65: Day 113: number analyzed (Participants) | 4 | 4
  CK-18/M65: Day 113 | 235.205 (290.846) | -188.638 (244.324)
  CK-18/M30: Day 29 | -24.282 (374.146) | -68.896 (96.850)
  CK-18/M30: Day 57 | 7.530 (445.509) | -20.074 (219.782)
  CK-18/M30: Day 85 | -54.988 (315.261) | -81.492 (271.506)
  CK-18/M30: Day 113: number analyzed (Participants) | 4 | 4
  CK-18/M30: Day 113 | 146.412 (273.673) | -170.793 (235.722)

9. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Ferritin at Days 29, 57, 85, and 113
Description: as for outcome 7
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
micrograms per liter (mcg/L)
  Day 29 | 6.4 (12.0) | 10.8 (25.9)
  Day 57 | 19.4 (23.5) | 3.6 (15.6)
  Day 85 | 11.8 (16.6) | -4.0 (2.4)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 6.0 (5.7) | -12.8 (11.1)

10. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Fibroblast Growth Factor 19 and Fibroblast Growth Factor 21 at Days 29, 57, 85, and 113
Description: as for outcome 7
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
picograms per milliliter (pg/mL)
  Fibroblast Growth Factor 19: Day 29 | -24.4 (80.6) | -42.8 (78.0)
  Fibroblast Growth Factor 19: Day 57 | -10.4 (51.2) | -18.8 (85.3)
  Fibroblast Growth Factor 19: Day 85 | 28.4 (77.5) | -13.0 (100.6)
  Fibroblast Growth Factor 19: Day 113: number analyzed (Participants) | 4 | 4
  Fibroblast Growth Factor 19: Day 113 | -7.8 (61.3) | -19.8 (35.3)
  Fibroblast Growth Factor 21: Day 29 | 9.98 (91.38) | 128.84 (171.50)
  Fibroblast Growth Factor 21: Day 57 | -36.36 (188.91) | 195.94 (315.73)
  Fibroblast Growth Factor 21: Day 85 | 120.68 (191.62) | 81.56 (130.68)
  Fibroblast Growth Factor 21: Day 113: number analyzed (Participants) | 4 | 4
  Fibroblast Growth Factor 21: Day 113 | 3.50 (291.41) | 56.35 (87.53)

11. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Hyaluronic Acid, Procollagen 3 N-Terminal Propeptide (PIIINP) and Tissue Inhibitor of Metalloproteinase 1 (TIMP1) at Days 29, 57, 85, and 113
Description: as for outcome 7
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
nanograms per milliliter (ng/mL)
  Hyaluronic Acid: Day 29 | -2.958 (11.689) | -8.800 (10.991)
  Hyaluronic Acid: Day 57 | -0.272 (9.228) | -3.654 (10.528)
  Hyaluronic Acid: Day 85 | 4.408 (16.612) | -3.518 (15.130)
  Hyaluronic Acid: Day 113: number analyzed (Participants) | 4 | 4
  Hyaluronic Acid: Day 113 | 1.592 (16.445) | -0.422 (19.347)
  Procollagen 3 N-Terminal Propeptide: Day 29 | -3.018 (14.079) | -2.878 (3.138)
  Procollagen 3 N-Terminal Propeptide: Day 57 | 1.730 (6.928) | -2.762 (3.242)
  Procollagen 3 N-Terminal Propeptide: Day 85 | -1.710 (6.730) | -0.470 (5.270)
  Procollagen 3 N-Terminal Propeptide: Day 113: number analyzed (Participants) | 4 | 4
  Procollagen 3 N-Terminal Propeptide: Day 113 | -7.015 (11.902) | -0.530 (3.701)
  Tissue Inhibitor of Metalloproteinase 1: Day 29 | -3.56 (25.38) | -8.52 (8.98)
  Tissue Inhibitor of Metalloproteinase 1: Day 57 | 2.80 (15.35) | -26.20 (32.29)
  Tissue Inhibitor of Metalloproteinase 1: Day 85 | 16.02 (24.84) | -26.26 (25.43)
  Tissue Inhibitor of Metalloproteinase 1: Day 113: number analyzed (Participants) | 4 | 4
  Tissue Inhibitor of Metalloproteinase 1: Day 113 | 10.92 (21.58) | -31.35 (37.95)

12. Secondary Outcome: Pharmacodynamics - Other Liver Markers: Change From Baseline in Alpha-2 Macroglobulin at Days 29, 57, 85, and 113
Description: as for outcome 7
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
gram per liter (g/L)
  Day 29 | -0.098 (0.254) | -0.282 (0.133)
  Day 57 | 0.124 (0.213) | -0.118 (0.064)
  Day 85 | -0.030 (0.328) | -0.204 (0.129)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | -0.105 (0.319) | -0.037 (0.157)

13. Secondary Outcome: Pharmacodynamics - Glucose Homeostasis Markers: Change From Baseline in Fasting Plasma Glucose (FPG) at Days 15, 29, 57, 85, and 113
Description: Blood samples were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
millimoles per liter (mmol/L)
  Day 15 | 0.22 (0.34) | 0.22 (0.28)
  Day 29 | 0.34 (0.61) | 0.12 (0.47)
  Day 57: number analyzed (Participants) | 5 | 4
  Day 57 | 0.18 (0.58) | 0.10 (0.24)
  Day 85 | 0.28 (0.63) | 0.08 (0.45)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.58 (0.52) | 0.17 (0.35)

14. Secondary Outcome: Pharmacodynamics - Glucose Homeostasis Markers: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Days 15, 29, 57, 85, and 113
Description: HOMA IR measures insulin resistance based on fasting glucose and insulin measurements: HOMA IR = fasting plasma insulin (micro international units per milliliter [mcIU/mL]) * fasting plasma glucose (mmol/L) / 22.5. A higher value indicates a greater insulin resistance. Blood samples were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Insulin resistance
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Insulin resistance
  Day 15 | 10.720 (17.650) | -3.640 (5.215)
  Day 29 | 16.498 (43.577) | -4.028 (6.512)
  Day 57: number analyzed (Participants) | 5 | 4
  Day 57 | 4.958 (15.472) | -5.448 (3.572)
  Day 85 | 3.742 (6.853) | -1.968 (7.112)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 13.323 (22.795) | -4.623 (6.883)

15. Secondary Outcome: Pharmacodynamics - Glucose Homeostasis Markers: Change From Baseline in Fasting Insulin at Days 15, 29, 57, 85, and 113
Description: Blood samples were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1. Here, "mIU/L" was abbreviated as "milli-international unit per liter".
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mIU/L
  Day 15 | 30.88 (53.53) | -15.66 (20.92)
  Day 29 | 40.12 (116.20) | -16.76 (24.12)
  Day 57: number analyzed (Participants) | 5 | 4
  Day 57 | 12.42 (41.76) | -23.10 (12.58)
  Day 85 | 9.70 (15.49) | -7.48 (26.76)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 34.15 (58.20) | -19.57 (25.56)

16. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Total Cholesterol (TC) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | -0.070 (0.440) | -0.328 (0.230)
  Day 29 | -0.356 (0.252) | -0.288 (0.347)
  Day 57 | 0.380 (0.565) | -0.286 (0.129)
  Day 85 | 0.298 (0.836) | -0.274 (0.306)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.665 (0.919) | 0.105 (0.270)

17. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Non High-density Lipoprotein Cholesterol (Non-HDL-C) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | -0.134 (0.414) | -0.348 (0.163)
  Day 29 | -0.324 (0.196) | -0.316 (0.432)
  Day 57 | 0.368 (0.340) | -0.316 (0.194)
  Day 85 | 0.156 (0.615) | -0.420 (0.290)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.605 (0.714) | -0.038 (0.229)

18. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum High-density Lipoprotein Cholesterol (HDL-C) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | 0.060 (0.068) | 0.020 (0.223)
  Day 29 | -0.032 (0.124) | 0.032 (0.137)
  Day 57 | 0.008 (0.228) | 0.030 (0.168)
  Day 85 | 0.138 (0.278) | 0.150 (0.191)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.065 (0.259) | 0.150 (0.047)

19. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Low-density Lipoprotein (LDL-C) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: Analysis was performed on ITT population. Here, 'number analyzed' signifies participants who were evaluable for this outcome measure at the specific time points.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | -0.224 (0.365) | -0.084 (0.213)
  Day 29 | -0.344 (0.184) | -0.076 (0.355)
  Day 57 | 0.314 (0.355) | -0.038 (0.078)
  Day 85 | 0.080 (0.686) | -0.184 (0.223)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.385 (0.691) | 0.108 (0.134)

20. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Triglycerides at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | 0.200 (0.363) | -0.576 (0.442)
  Day 29 | 0.042 (0.214) | -0.530 (0.385)
  Day 57 | 0.124 (0.326) | -0.606 (0.384)
  Day 85 | 0.170 (0.389) | -0.532 (0.399)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.485 (0.918) | -0.315 (0.353)

21. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Calculated Very Low-density Lipoprotein Cholesterol (VLDL-C) at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
mmol/L
  Day 15 | 0.086 (0.172) | -0.270 (0.200)
  Day 29 | 0.018 (0.103) | -0.244 (0.168)
  Day 57 | 0.052 (0.140) | -0.282 (0.176)
  Day 85 | 0.072 (0.168) | -0.240 (0.176)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.215 (0.419) | -0.153 (0.156)

22. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Apolipoprotein A-1 at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
grams per liter (g/L)
  Day 15 | 0.112 (0.129) | -0.058 (0.149)
  Day 29 | 0.012 (0.139) | -0.058 (0.144)
  Day 57 | 0.108 (0.211) | -0.060 (0.176)
  Day 85 | 0.128 (0.268) | 0.016 (0.160)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.103 (0.313) | 0.048 (0.060)

23. Secondary Outcome: Pharmacodynamics - Serum Lipid Parameters: Change From Baseline in Serum Apolipoprotein B at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
g/L
  Day 15 | -0.058 (0.064) | -0.082 (0.074)
  Day 29 | -0.098 (0.081) | -0.078 (0.097)
  Day 57 | 0.066 (0.092) | -0.062 (0.086)
  Day 85 | 0.020 (0.189) | -0.036 (0.090)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.117 (0.209) | -0.005 (0.135)

24. Secondary Outcome: Pharmacodynamics - Change From Baseline in Body Weight at Days 15, 29, 57, 85, and 113
Description: Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
kilograms (kg)
  Day 15 | -0.08 (3.03) | -0.92 (1.70)
  Day 29 | -0.32 (4.54) | -0.98 (2.06)
  Day 57 | 0.73 (5.18) | -0.68 (3.27)
  Day 85 | 1.54 (5.42) | 0.24 (4.07)
  Day 113: number analyzed (Participants) | 4 | 5
  Day 113 | 4.40 (3.05) | 0.73 (4.63)

25. Secondary Outcome: Pharmacodynamics - Change From Baseline in Body Mass Index (BMI) Z-Score at Days 15, 29, 57, 85, and 113
Description: The BMI for a given age (in years) and gender (male) was converted to an exact z-score. Given a participant's age, sex, BMI, and an appropriate reference standard, a BMI Z-score was determined. BMI Z-score >=85th percentile was considered as overweight. Z-score was a statistical measure to describe whether a mean was above or below the standard. A Z-score of 0 was equal to the mean and is considered normal. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. Negative values are indicative of decrease in BMI (weight loss) and positive values are indicative of increase in BMI. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Z-Score
  Day 15 | -0.064 (0.146) | -0.054 (0.095)
  Day 29 | -0.091 (0.247) | -0.054 (0.110)
  Day 57 | -0.108 (0.284) | -0.058 (0.162)
  Day 85 | -0.074 (0.290) | -0.026 (0.197)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.068 (0.116) | 0.022 (0.247)

26. Secondary Outcome: Pharmacodynamics - Change From Baseline in Waist Circumference at Days 15, 29, 57, 85, and 113
Description: Waist circumference (in centimeters [cm]) was measured at the midpoint between the lower margin of the least palpable rib and the top of the iliac crest. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
cm
  Day 15 | -1.056 (2.953) | -0.998 (2.961)
  Day 29 | -0.656 (3.654) | -2.010 (2.625)
  Day 57 | -0.316 (3.520) | -2.054 (4.106)
  Day 85 | 0.252 (3.379) | -1.346 (3.894)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 1.625 (2.394) | -0.580 (4.099)

27. Secondary Outcome: Pharmacodynamics - Inflammatory Marker: Change From Baseline in Fibrinogen at Days 29, 57, 85, and 113
Description: Blood samples to assess fibrinogen levels were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
micromoles per liter (mcmol/L)
  Day 29 | -1.450 (1.265) | -2.474 (1.418)
  Day 57 | -0.524 (1.309) | -2.220 (0.756)
  Day 85 | -1.340 (1.492) | -1.748 (1.000)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | -0.295 (1.936) | -1.150 (1.841)

28. Secondary Outcome: Pharmacodynamics - Inflammatory Marker: Change From Baseline in Haptoglobin at Days 29, 57, 85, and 113
Description: Blood samples to assess Haptoglobin level were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
g/L
  Day 29 | -0.086 (0.102) | -0.350 (0.244)
  Day 57 | 0.068 (0.118) | -0.300 (0.209)
  Day 85 | 0.066 (0.077) | -0.298 (0.236)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.178 (0.208) | -0.058 (0.081)

29. Secondary Outcome: Pharmacodynamics - Inflammatory Marker: Change From Baseline in Interleukin-6 at Days 29, 57, 85, and 113
Description: Blood samples to assess Interleukin-6 level were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
picograms per milliliter (pg/mL)
  Day 29 | 0.036 (0.080) | 0.142 (0.751)
  Day 57 | 0.100 (0.224) | -0.092 (1.096)
  Day 85 | 0.142 (0.243) | 0.062 (0.809)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.143 (0.285) | 0.078 (0.534)

30. Secondary Outcome: Pharmacodynamics - Inflammatory Marker: Change From Baseline in Tumor Necrosis Factor Alpha at Days 29, 57, 85, and 113
Description: Blood samples to assess Necrosis Factor Alpha level were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
pg/mL
  Day 29 | -0.134 (0.437) | -0.460 (0.857)
  Day 57 | 0.068 (0.388) | -0.270 (0.651)
  Day 85 | -0.068 (0.416) | -0.622 (0.939)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 0.163 (0.534) | -0.445 (0.988)

31. Secondary Outcome: Pharmacodynamics - Inflammatory Marker: Change From Baseline in Plasminogen Activator Inhibitor-1 at Days 29, 57, 85, and 113
Description: Blood samples to assess plasminogen activator inhibitor-1 level were taken after minimum 10 hours of fasting. Baseline was defined as the last measurement before first intake of study treatment on Day 1. Here, "IU/mL" was abbreviated as International units per milliliter.
Time Frame: Baseline (Day 1), Day 29, 57, 85, and 113
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
IU/mL
  Day 29: number analyzed (Participants) | 4 | 5
  Day 29 | -8.95 (14.19) | -1.40 (10.33)
  Day 57: number analyzed (Participants) | 4 | 5
  Day 57 | 9.68 (32.87) | 2.46 (15.03)
  Day 85: number analyzed (Participants) | 4 | 5
  Day 85 | -2.43 (7.57) | 2.62 (23.77)
  Day 113: number analyzed (Participants) | 4 | 4
  Day 113 | 5.75 (26.71) | 5.40 (5.42)

32. Secondary Outcome: Pharmacodynamics - Change From Baseline in Pediatric Quality of Life (PedsQL™) (Version 4.0) Generic Core Scales at Day 85
Description: The child, adolescent and parent/legal guardian PedsQL™ (Version 4.0) generic core scales was used to measure health-related quality of life (HRQOL). The response information was completed by the participant and by a parent/legal guardian individually. It consisted of 23 item questionnaire encompassing 4 core scale domains: Physical Functioning (8 items); Emotional Functioning (5 items); Social Functioning (5 items); and School Functioning (5 items). Items were scored on a 5 point Likert-type response scale: 0=never a problem to 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). Once scored, items were reverse scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), where higher scores indicated better HRQOL. Total Scale Score was the sum of all the items over the number of items answered on all the Scales. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
units on a scale
  Parent: number analyzed (Participants) | 4 | 5
  Parent | -3.80 (13.76) | -13.04 (11.32)
  Participants | -3.04 (1.42) | -3.04 (9.01)

33. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical in a participant or clinical investigation patient administered a pharmaceutical (investigational) product and which does not necessarily have to have a causal relationship with this treatment. A Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was another medically important condition. TEAEs were defined as AEs that started prior to first study drug dose and that worsened after, and the AEs that started on or after first study drug dose. TEAEs: Serious and non-serious AEs.
Time Frame: From Screening visit (signature of informed consent) up to last dose of study drug + 30 days (i.e., up to Day 113)
Population: Analysis was performed safety population that included participants who had received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Participants with TEAEs | 2 | 0
  Participants with Serious TEAEs | 0 | 0

34. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) Measurement
Description: ECG measurements were taken with the participants in resting position for at least 10 minutes. The investigator determined whether abnormal assessment results were clinically significant or not. The number of participants with abnormal clinically significant ECG findings were reported. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Day 85
Population: Analysis was performed safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Baseline (Day1): Abnormal, clinically significant | 0 | 0
  Day 85: Abnormal, clinically significant | 0 | 0

35. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: Fasting blood samples (collected after 10 hours fasting) were used to assess the following clinical chemistry parameters: creatinine, glomerular filtration rate, creatinine clearance, total proteins, albumin, electrolytes (sodium, potassium, chloride, calcium), uric acid, urea nitrogen, urea, creatine phosphokinase (CPK), AST, ALT, GGT, ALP, total and conjugated bilirubin, high sensitivity C-reactive protein, fasting plasma glucose, fasting insulin, HOMA-IR, fructosamine, C-peptide, free fatty acids, glycated hemoglobin A1c, cystatin C. Abnormal clinical chemistry values were classified based on reference range: lower limit of normality (LLN); normal (>= LLN and <= upper limit of normality [ULN]); > ULN and <3 ULN; >=3 ULN and <5 ULN and >=5 ULN. Only the parameters for which at least one value of abnormality were reported and presented in this outcome measure.
Time Frame: At Day 85 (i.e., end of treatment)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Total proteins: >ULN and <3 ULN | 1 | 1
  Albumin: >ULN and <3 ULN | 1 | 0
  CPK: >ULN and <3 ULN | 0 | 1
  AST: >ULN and <3 ULN | 3 | 0
  ALT: >ULN and <3 ULN | 3 | 4
  ALT: >=3 ULN and <5 ULN | 1 | 0
  ALT: >=5 ULN | 1 | 0
  GGT: >ULN and <3 ULN | 2 | 2
  GGT: >=3 ULN and <5 ULN | 1 | 0
  GGT: >=5 ULN | 1 | 0
  ALP: >ULN and <3 ULN | 1 | 0
  Total Bilirubin: >ULN and <3 ULN | 0 | 1
  Conjugated Bilirubin: >ULN and <3 ULN | 0 | 1
  C Reactive Protein: >ULN and <3 ULN | 0 | 1
  Fasting plasma glucose: >ULN and <3 ULN | 1 | 0
  Fasting insulin: >ULN and <3 ULN | 3 | 5
  Fasting insulin: >=3 ULN and <5 ULN | 2 | 0
  C-peptide: >ULN and <3 ULN | 4 | 2
  Hemoglobin A1C: >ULN and <3 ULN | 1 | 0

36. Secondary Outcome: Number of Participants With Abnormal Hematology and Coagulation Parameters
Description: Fasting blood samples (collected after 10 hours fasting) were used to assess the following hematology and coagulation parameters: hemoglobin, hematocrit, red blood cells (RBC), white blood cells (WBC), neutrophils, eosinophils, basophils, lymphocytes, monocytes, platelets, prothrombin time (PT) and international normalized ratio (INR). Hematology and coagulation values were classified based on the reference range: LLN; normal (>= LLN and <= ULN); > ULN and <3 ULN; >=3 ULN and <5 ULN and >=5 ULN.
Time Frame: At Day 85 (i.e., end of treatment)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Haemoglobin: >ULN and <3 ULN | 0 | 0
  Hematocrit: >ULN and <3 ULN | 0 | 0
  RBC: >ULN and <3 ULN | 0 | 1
  WBC: >ULN and <3 ULN | 0 | 0
  Neutrophils: >ULN and <3 ULN | 0 | 0
  Eosinophils: >ULN and <3 ULN | 0 | 0
  Basophils: >ULN and <3 ULN | 0 | 0
  Lymphocytes: >ULN and <3 ULN | 0 | 0
  Monocytes: >ULN and <3 ULN | 0 | 0
  Platelets: >ULN and <3 ULN | 0 | 0
  PT: >ULN and <3 ULN | 0 | 0
  INR: >ULN and <3 ULN | 0 | 0

37. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters
Description: Blood samples were collected to assess the following urinalysis parameters: alpha-1 macroglobulin, N-acetyl glucosamide, neutrophil gelatinase-associated lipocalin, albumin, and creatinine. Abnormal urinalysis values were classified based on the reference range: LLN; normal (>= LLN and <= ULN); > ULN and <3 ULN; >=3 ULN and <5 ULN and >=5 ULN.
Time Frame: At Day 85 (i.e., end of treatment)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Alpha-1 Microglobulin: >ULN and <3 ULN | 0 | 0
  N-Acetyl Glucosamide: >ULN and <3 ULN | 0 | 0
  Neutrophil Gelatinase-associated: >ULN and <3 ULN | 0 | 0
  Albumin: : >ULN and <3 ULN | 0 | 0
  Creatinine | 0 | 0

38. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs were taken before any invasive procedures. Following vital signs were assessed: systolic blood pressure, diastolic blood pressure, heart rate. Abnormal vita signs was defined as any abnormal findings in the vital sign parameters and were categorized as 'abnormal, not clinically significant (NCS)' and 'abnormal, clinically significant (CS)'.
Time Frame: At Day 85 (i.e., end of treatment)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 5 | 5
Participants
  Systolic Blood Pressure:Abnormal, not clinically significant | 0 | 0
  Systolic Blood Pressure: Abnormal, clinically significant | 0 | 0
  Diastolic Blood Pressure: Abnormal, not clinically significant | 0 | 0
  Diastolic Blood Pressure: Abnormal, clinically significant | 0 | 0
  Heart Rate: Abnormal, not clinically significant | 0 | 0
  Heart Rate: Abnormal, clinically significant | 0 | 0

39. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination at Baseline, Days 15, 29, 57, 85, and 113
Description: Physical examination findings were collected according to pre-defined body systems: general appearance; skin; eyes; ears; nose; throat; neck and thyroid; lungs; heart; upper/lower extremities; lymph nodes; abdomen; musculoskeletal system; basic neurological assessment. Additional systems were evaluated as needed. Clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care. Participants with at least one clinically significant abnormality in physical examination were reported and presented in this outcome measure. Baseline was defined as the last measurement before first intake of study treatment on Day 1.
Time Frame: Baseline (Day 1), Days 15, 29, 57, 85, and 113
Population: Analysis was performed on safety population. Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
Number analyzed (Participants) | 4 | 2
Participants
  Baseline (Day 1) | 4 | 2
  Day 15 | 0 | 0
  Day 29 | 1 | 0
  Day 57 | 0 | 0
  Day 85 | 0 | 0
  Day 113 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from screening through 30 days after last dose of study drug (i.e., up to Day 113) regardless of seriousness or relationship to study drug.
Description: Reported AEs were TEAEs that started prior to first study drug dose and that worsened after, and the AEs that started on or after first study drug dose. Analysis was performed on safety population.
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elafibranor 80 mg (N=5) | Elafibranor 120 mg (N=5)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to lack of efficacy (but not due to safety) in a Phase 3 trial of elafibranor in adult participants with NASH and fibrosis, this study in pediatric NASH was prematurely terminated. Therefore, participants >=12 to <=17 years of age were only involved in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor retains exclusive ownership of all data, results, reports, findings, discoveries, and any other information collected during this study; these may not be published, given, or disclosed, either in part or in whole, by the Investigator or by any person under his/her authority to any third party without the prior express consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03883607/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03883607/SAP_001.pdf